CLINICAL TRIAL: NCT01237600
Title: Efficacy of Cultivated Corneal Epithelial Stem Cell for Ocular Surface Reconstruction
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Pinnita Prabhasawat, Associate Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 447/2550(EC2)
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Severe Ocular Surface Damage; Limbal Deficiency
Keywords: Ocular surface damage; Limbal deficiency; Cultivated corneal epithelial stem cell transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cultivated limbal transplantation (Experimental)
  Interventions: Procedure: Cultivated limbal transplantation

INTERVENTIONS:
Procedure: Cultivated limbal transplantation — Cultivated corneal epithelial stem cell transplantation. Autograft, Living related allograft, and Cadaveric allograft

SUMMARY:
The purpose of this study is to elucidate the appropriate condition of developing cultivated corneal epithelial graft and evaluate the surgical outcome of transplantation of the cultivated corneal epithelial stem cell in the patients.

DETAILED DESCRIPTION:
Ocular surface damage caused by severe ocular surface diseases, particularly thermal and chemical burn or Stevens-Johnson syndrome result in corneal epithelial defect, corneal vascularization, corneal conjunctivalization and loss of transparency. Corneal limbal stem cell transplantation has been demonstrated to improve the outcome of ocular surface reconstruction. However, the conventional management of allograft limbal transplantation generally has unsatisfactory outcome because of high risk of rejection and requires long-life immunosuppressive medications.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral/Bilateral limbal stem cell deficiency proved by specific clinical features and impression cytology result

Exclusion Criteria:

* Age under 18
* Active ocular infection, Severe dry eye, Uncontrolled glaucoma
* Immunocompromised host
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-01; Primary Completion 2011-04 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Ocular surface status (signs of limbal deficiency and immunopathological markers) | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Pinnita Prabhasawat, MD, Principal Investigator — Mahidol University
Locations (1):
- Pinnita Prabhasawat, MD, Bangkok, Thailand